CLINICAL TRIAL: NCT02943291
Title: Adipose Tissue Function and Response to Exercise Training in Women With and Without Polycystic Ovary Syndrome
Acronym: HIT-FAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Liverpool John Moores University (Other); Australian Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/545
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Exercise therapy; Adipose tissue; Mitochondria; Oxidative Phosphorylation
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — High-Intensity Interval Training; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4x4 minutes interval training (Experimental): 4x4 minutes high intensity interval training with 4 minute intervals
  Interventions: Behavioral: 4x4 minutes high intensity interval training
- 10x1 minute interval training (Experimental): 10x1 minute high intensity interval training with 1 minute intervals
  Interventions: Behavioral: 10x1 minute high intensity interval training

INTERVENTIONS:
Behavioral: 4x4 minutes high intensity interval training — Treadmill running/walking with 10 minutes warm-up at 60-70% of maximum heart rate, 4x4 minute intervals at 90-95% of maximum heart rate separated by 3-minutes active pauses at 60-70% of maximum heart rate, and 3 minutes cool-down.
  Other Names: High-intensity exercise; Aerobic exercise
  Arms: 4x4 minutes interval training
Behavioral: 10x1 minute high intensity interval training — Treadmill running/walking with 10 minutes warm-up at 60-70% of maximum heart rate, ten 1-minute intervals at maximal intensity (that can be performed for one minute), separated by 1-minutes active pauses at 60-70% of maximum heart rate, and 3 minutes cool-down.
  Other Names: High-intensity exercise; Aerobic exercise
  Arms: 10x1 minute interval training

SUMMARY:
The primary aim of this trial is to investigate adipose tissue function in women with and without polycystic ovary syndrome (PCOS). PCOS is a common endocrine disorder in young women. The pathogenesis behind PCOS is complex and only partly understood, and deeper mechanistic insight is needed. Insulin resistance is a central feature of PCOS, and recent studies have suggested that this is linked to aberrant adipose tissue function. Exercise training has been found to improve the symptoms in PCOS, but we need more knowledge about why. While processes involved in skeletal muscle oxidative remodeling are well described, it is to a large extent unknown whether the oxidative capacity of human adipose tissue is modified by endurance training. The women included in this study will be matched (for body mass index, body weight, and age) to participants in another study. This will enable the investigators to do a comparison between cases (women with PCOS) and controls (women without PCOS) at baseline, and to assess the responses to exercise training in adipose tissue.

ELIGIBILITY:
Inclusion Criteria:

* eumenorrheic
* matching PCOC group in IMPROV-IT study (NCT02419482)
* Living nearby St Olavs Hospital, Trondheim, Norway

Exclusion Criteria:

* Signs of hyperandrogenism
* Regular high intensity endurance (two or more times per week of vigorous exercise).
* Concurrent treatments (insulin sensitizers or drugs known to affect gonadotropin or ovulation, with a wash out period of 1 months prior to inclusion).
* On-going pregnancy
* Hormonal contraception
* Breastfeeding within 24 weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
mitochondrial oxidative phosphorylation capacity | 16 weeks
  assessed with high resolution respirometry
production of reactive oxygen species | 16 weeks
  assessed with high resolution respirometry

SECONDARY OUTCOMES:
Adipokine secretion | 16 weeks
lipid droplet size in adipocytes | 16 weeks
Whole-body fat oxydation rate | 16 weeks
Insulin sensitivity | 16 weeks
  2h oral glucose tolerance test (OGGT)
Whole-body peak oxygen uptake | 16 weeks
Adipokine gene expression | 16 weeks
Total protein abundance in adipose tissue | 16 weeks
  quantified using standard Western Blot method
"blood markers of cardiometabolic health" | 16 weeks
Body composition | 16 weeks
  assessed by impedance scale (InBody)
blood pressure | 16 weeks
endothelial function | 16 weeks
  measured by flow-mediated dilatation of the brachial artery
Intima media thickness | 16 weeks
  measured by ultrasound
Total cholesterol in blood | 16 weeks
HDL cholesterol in blood | 16 weeks
LDL cholesterol in blood | 16 weeks
blood glucose | 16 weeks
blood insulin | 16 weeks
Glycosylated Hemoglobin (HbA1c) in blood | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn L Helbostad, phd prof, Study Director — Norwegian University of Science and Technology
Locations (2):
- Centre of Exercise and Nutrition, Mary MacKillop Institute for Health Research, AUC, Melbourne, Australia
- Department of circulation and medical imaging , NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lionett S, Kiel IA, Camera DM, Vanky E, Parr EB, Lydersen S, Hawley JA, Moholdt T. Circulating and Adipose Tissue miRNAs in Women With Polycystic Ovary Syndrome and Responses to High-Intensity Interval Training. Front Physiol. 2020 Jul 30;11:904. doi: 10.3389/fphys.2020.00904. eCollection 2020. PMID 32848854
- [Result] Kiel IA, Jones H, Lionett S, Rosbjorgen R, Lydersen S, Vanky E, Moholdt T. Cardiovascular Health Does Not Change Following High-Intensity Interval Training in Women with Polycystic Ovary Syndrome. J Clin Med. 2022 Mar 15;11(6):1626. doi: 10.3390/jcm11061626. PMID 35329952
- [Result] Lionett S, Kiel IA, Rosbjorgen R, Lydersen S, Larsen S, Moholdt T. Absent Exercise-Induced Improvements in Fat Oxidation in Women With Polycystic Ovary Syndrome After High-Intensity Interval Training. Front Physiol. 2021 Mar 24;12:649794. doi: 10.3389/fphys.2021.649794. eCollection 2021. PMID 33841184